CLINICAL TRIAL: NCT03145506
Title: Spectrally Guided Mohs Surgery
Status: Completed | Type: Observational
Sponsor: Seton Healthcare Family (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: CR-15-117
Record Dates: First submitted 2017-04-24; First posted 2017-05-09 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mohs Surgery Patients: Adult patients undergoing Mohs surgery for treatment of BCC or SCC
  Interventions: Device: Multimodal Spectroscopy

INTERVENTIONS:
Device: Multimodal Spectroscopy — optical measurement of excised tissue

SUMMARY:
Freshly excised or freshly frozen tissue for Raman analysis will be obtained from a dermatology practice affiliated with UMCB. In the course of the routine removal of benign or malignant tumors in the office, skin cancer surgeons routinely check frozen sections to ensure adequate margins are obtained. Consent will be obtained from patients to provide freshly excised or freshly frozen leftover tissue obtained during Mohs surgery to be discarded after histological diagnosis. Freshly excised tissue will be measured at the time of excision before processing, while the freshly frozen tissue samples will be stored in a freezer at the Mohs clinic and transferred to the UT- Austin campus for spectroscopic analysis.

DETAILED DESCRIPTION:
The current standard-of-care in the identification of skin cancer is visual inspection followed by biopsy and histopathology of suspicious skin sites. Since a physician is required to perform this biopsy, there is often a delay in diagnosis, resulting in deeper, more aggressive tumors and increased mortality from malignant melanoma (MM). Therefore, a non-invasive method to inspect these lesions would be of great clinical importance.

An initial prototype of a noninvasive diagnostic device was developed based on optical spectroscopy and completed a clinical study in 76 patients that demonstrated high diagnostic accuracy for the detection of skin cancer (IRB # CR-10-004). This initial prototype consisted of two separate devices and probes: one to collect Raman spectra (RS) and the other to collect diffuse reflectance and laser induced fluorescence spectra (DRS+LIFS). type, but a combination of modalities gave the best diagnostic performance for all types of skin cancer.

The addition of Raman spectroscopy improved diagnostic performance for both melanoma and non-melanoma skin cancer. However, the operation of the integrated systems was still conducted via two optical fiber probes (the first one for fluorescence and reflectance spectroscopy, the second one for Raman spectroscopy). The need to take measurements of the same lesion using two probes increased acquisition time, and the possible sampling site error. Recently, a device was developed that combined fiber optic probe that is capable for spectral acquisition of Raman, white light reflectance and laser induced fluorescence spectroscopy. Using this probe, acquisition time and sampling site error should be reduced. There is no significant difference in terms of performance between the previous two probes and the new probe.

Models have been developed to analyze reflectance and fluorescence spectroscopy data. In order to interpret Raman spectroscopy data in physiologically relevant parameters, a biophysical model needs to be developed. Similar models have been developed by other research groups for other types of tissue.

This study proposes to use the new technique of biophysical modeling to analyze our Raman spectra. At the core of the technique is the measurement of a set of "basis spectra" which are fit to the data using ordinary least-squares. Recently, biophysical models have been developed for atherosclerosis and breast cancer with very impressive diagnostic results, achieving 94% sensitivity and 96% specificity for breast cancer and 94% accuracy for atherosclerosis disease classification.

Raman microspectrometry will be used to measure basis spectra from various skin constituents. In this technique, Raman spectra are measured from freshly frozen tissue samples that are sliced into thin sections as is done in histology. A microscope system is used to focus the excitation laser beam to a small spot of approximately 2 mm in diameter on the sample, and a Raman spectrometer measures the emitted Raman spectrum. In this way, Raman spectra of individual microscopic tissue components can be isolated. These individual component spectra will be determined for keratin, cell nuclei, collagen, cytoplasm, melanin, water, sebaceous glands, etc.

ELIGIBILITY:
Inclusion Criteria:

* All individuals over 18 undergoing Mohs surgery for treatment of BCC or SCC

Exclusion Criteria:

* Under 18 years old, not undergoing Mohs surgery for treatment of BCC or SCC

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing treatment for SCC or BCC in local Mohs surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of spectroscopic device | 1 year
  comparison of spectroscopic data to frozen section pathology used in Mohs surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jason Reichenberg, MD, Principal Investigator — Seton Healthcare Family

IPD SHARING:
Plan to Share IPD: No